CLINICAL TRIAL: NCT05040516
Title: The Role of Selenoprotein Activity and Blood Renalase Level in the Pathogenesis of Hypertension and Obstructive Sleep Apnea
Brief Title: Selenoprotein and Renalase Blood Levels in Patients With Hypertensive Heart Disease and Obstructive Sleep Apnea
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Wroclaw Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: KB-39/2020
Record Dates: First submitted 2021-08-09; First posted 2021-09-10 (Actual); Last update posted 2021-09-10 (Actual); Status verified 2021-08

CONDITIONS: Hypertension; Obstructive Sleep Apnea
Keywords: hypertension; renalase; selenoprotein
MeSH Terms: conditions — Hypertension; Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Days
Biospecimen Retention: Samples With DNA — 10 ml of venous blood collected by venopuncture
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1: The planned procedures include: medical interview, physical examination with basic anthropometric measurements (age, height, body weight); biochemical tests including blood selenium, selenoproteins, renalase and creatinine levels; total antioxidant status (TAS), 24-hour Holter electrocardiography, polysomnography and echocardiography.
  A 10 ml of venous blood sample will be collected by venopuncture. Laboratory tests will be performed using commercially available standardized tests.

SUMMARY:
The aim of the study is to determine whether selenoprotein activity and blood renalase level correlate with subclinical hypertensive heart disease and obstructive sleep apnea. The correlation will be assessed using selected electrocardiographic, ultrasound and laboratory indicators.

DETAILED DESCRIPTION:
The study will be conducted in the Department and Clinic of Internal Medicine, Occupational Diseases, Hypertension and Clinical Oncology at Borowska 213 street in Wroclaw. This decision follows the high percentage of people with obstructive sleep apnea and hypertension among those hospitalized in the Clinic and also the wide availability of research tools in the hospital.

150 more patients with hypertension and obstructive sleep apnea will be included in the planned observational study.

The study is observational, research procedures are non-invasive and no additional medical experiment is planned. The study was approved by the Bioethics Committee of the Wroclaw Medical University.

Patients enrolled in the study will be asked to share the results of their previously performed examinations or, in case they do not have any, new examinations will be performed to complement the diagnostic process of hypertension and obstructive sleep apnea.

The planned procedures include: medical interview, physical examination with basic anthropometric measurements (age, height, body weight); biochemical tests including blood selenium, selenoproteins, renalase and creatinine levels; total antioxidant status (TAS), 24-hour Holter electrocardiography, polysomnography, ultrasound assessment of peripheral vascular endothelial function and echocardiography.

Laboratory tests will be performed using commercially available standardized tests. The levels of selenoproteins, renalase and creatinine in the blood, as well as TAS will be determined by ELISA (Enzyme-linked immunosorbent assay) in accordance with the instructions. Blood selenium level will be measured by means of atomic absorption spectrometry (AAS). 24-hour Holter ECG monitoring will be performed using a Lifecard CF recorder, followed by an analysis of the record by the Impresario Solo system (Delmar Reynolds, Hertford, UK). Ultrasound examination will be performed using the ProSound Alpha 6 (Aloka Inc, Tokyo, Japan).

ELIGIBILITY:
Inclusion Criteria:

* arterial hypertension

Exclusion Criteria:

* age <18
* pregnancy
* refusal to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study participants will be recruited among the patients of the Department of Internal and Occupational Diseases, Hypertension and Clinical Oncology in Wroclaw. 150 more consecutive patients with hypertension and obstructive sleep apnea will be included in the planned observational study.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2020-01-27 (Actual); Primary Completion 2021-10-01 (Estimated); Study Completion 2021-10-01 (Estimated)

PRIMARY OUTCOMES:
Assesment of blood renalase level | One day
  The Enzyme-linked immunosorbent assay (ELISA) to know blood renalase level
Assesment of blood selenoprotein P level | One day
  The Enzyme-linked immunosorbent assay (ELISA) to know blood selenoprotein P level
Assesment of the severity of obstructive sleep apnea | One day
  Full polysomnography
Assessment of arrhythmias | One day
  24-hour Holter ECG monitoring
Assessment of arrhythmias and cardiac morphology | One day
  Echocardiography

SECONDARY OUTCOMES:
Assesment of Blood Total Antioxidant Status (TAS) | One day
  The Enzyme-linked immunosorbent assay (ELISA) to know Blood Total Antioxidant Status (TAS)

CONTACTS AND LOCATIONS:
Overall Officials: Paweł Gać, ASSOC PROF, Study Chair — Wroclaw Medical University
Locations (1):
- Department of Hygiene, Wroclaw Medical University, Wroclaw, Lower Silesian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No